CLINICAL TRIAL: NCT02774499
Title: Preoperative Oral Methadone for Patients Undergoing Cardiac Surgery: Reduction of Postoperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, William McKay, MD FRCPC, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bio16-02
Record Dates: First submitted 2016-04-06; First posted 2016-05-17 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Experimental): Methadone 0.3 mg/kg (to a maximum of 30 mg) will be given to the patient preoperatively.
  Interventions: Drug: Methadone
- Placebo (Placebo Comparator): Equivalent volume (5mL) of syrup will be given to the patient preoperatively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methadone — 0.3mg/kg of methadone given preoperatively (to maximum of 30mg)
  Arms: Methadone
Drug: Placebo — equivalent volume (5mL) of syrup given preoperatively
  Arms: Placebo

SUMMARY:
Oral medications like gabapentin and acetaminophen are commonly given to patients prior to surgery to provide balanced anaesthesia. Intravenous methadone has been shown to decrease postoperative pain as well as postoperative nausea and vomiting, which are known barriers to discharge. Oral methadone would be a convenient alternative to give as a preoperative medication with its bioavailability approaching 80%. No clinical trials to date have explored the utility of oral methadone as a preoperative analgesic to improve postoperative outcomes. Current literature shows preoperative IV methadone reduces opioid consumption in the perioperative period for cardiac surgeries; therefore, investigators hypothesize that preoperative oral methadone will also reduce postoperative pain and opioid consumption in patients undergoing sternotomy for cardiac surgery.

DETAILED DESCRIPTION:
Investigators propose a prospective, randomized, double-blind, placebo-controlled trial to investigate the effects of preoperative oral methadone on postoperative pain. The trial will be conducted in compliance with the protocol, Good Clinical Practice (GCP), and University of Saskatchewan Research Ethics Committee principles using an intent-to-treat model. The primary endpoint will be postoperative pain in the ICU, and secondary outcomes will include morphine requirements as measured by Patient Controlled Analgesia (PCA). Secondary endpoints include opioid consumption at 15 minutes and at 2, 4, 8, 12, 24, 48, and 72 hours post extubation. Other secondary endpoints include the following: pain with cough (using a 0-10 verbal pain scale) measured at the time of extubation then daily until post-op day three. Secondary outcomes that will be recorded from nursing assessment records include: incidence of nausea and/or vomiting requiring antiemetics, pruritus, hypoventilation (respiratory rate less than 8 breaths/min), hypoxemia (oxygen saturation less than 90%), time to extubation, and sedation (Richmond Agitation-Sedation Scale of -4 or -5).

Patients will receive a dose of either oral methadone or placebo prior to entering the operating room. The dose given will be 0.3 mg/kg (to a maximum of 30 mg) or equivalent volume of placebo. An blinded research assistant will receive an envelope the morning of surgery outlining if the patient is in group A or B as well as their weight in kg. For the methadone arm the research assistant will prepare the appropriate amount of methadone, which is dispensed as 10 mg/mL, and dilute it to a total volume of 5 mL in sugary syrup to mask its taste. For the placebo arm a similar volume will be mixed at a 0.3 mg/kg volume and diluted to a total volume of 5 mL of sugary syrup. The methadone or placebo will be given to the researcher in a syringe. The researcher will give syringe to the patient and the patient will administer the solution to themself orally prior to entering the operating room.

ELIGIBILITY:
Inclusion Criteria:

* presenting for elective first-time CABG cardiac surgery with anticipated extubation within 12 hours

Exclusion Criteria:

* < 18 years of age
* preoperative renal failure requiring dialysis or serum creatinine greater than 176 µmol/L
* significant hepatic dysfunction (liver function tests more than twice the upper limit of normal)
* ejection fraction less than 30%
* corrected QT interval (QTc) on ECG > 440ms for men and 450ms for women
* pulmonary disease necessitating home oxygen therapy
* preoperative requirement for inotropic agents or intra-aortic balloon pump to maintain hemodynamic stability
* emergency surgery
* allergy to methadone
* use of preoperative opioids or recent history of opioid abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pain score (VRS) | 24 hours
  Pain score as measured by 0-10 Verbal Rating Score (VRS)

SECONDARY OUTCOMES:
Total Morphine Consumption (mg) | 72 hours
  Total dose in mg of IV morphine administered via Patient Controlled Analgesia
Pain score (VRS) | Up to 72 hours postoperative
  Pain score as measured by 0-10 Verbal Rating Score (VRS)
Time to extubation | up to 24 hours postoperative
  Time from start of surgery until removal of endotracheal tube in ICU
Level of sedation | up to 72 hours postoperative
  Level of sedation as measured by the Richmond Agitation-Sedation Scale (RASS) in ICU
Incidence of opioid-related side effects | up to 72 hours postoperative
  Incidence of as nausea, vomiting, pruritus, hypoventilation, and hypoxia during a seventy-two hour monitoring period

CONTACTS AND LOCATIONS:
Overall Officials: William PS McKay, MD FRCPC, Principal Investigator — Department of Anesthesiology, University of Saskatchewan
Locations (1):
- Saskatoon Health Region, 410 22nd Street East, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bolton TM, Chomicki SO, McKay WP, Pikaluk DR, Betcher JG, Tsang JC. Preoperative oral methadone for postoperative pain in patients undergoing cardiac surgery: A randomized double-blind placebo-controlled pilot. Can J Pain. 2019 Apr 9;3(1):49-57. doi: 10.1080/24740527.2019.1575695. eCollection 2019. PMID 35005393